CLINICAL TRIAL: NCT01289574
Title: Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Clinical Study to Evaluate the Safety and Efficacy of 0.1% and 0.025% ASC-J9 Creams Applied Topically Twice Daily for 12 Weeks for the Treatment of Facial Acne Vulgaris
Brief Title: Topical ASC-J9 Cream for Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AndroScience Corp (Industry)
Collaborators: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC-J9-202
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Acne
Keywords: androgen receptor degradation enhancer
MeSH Terms: conditions — Acne Vulgaris | interventions — 1,7-bis(4-hydroxy-3-methoxyphenyl)-1,4,6-heptatrien-3-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle control cream (Placebo Comparator)
  Interventions: Drug: ASC-J9
- 0.025% ASC-J9 cream (Experimental)
  Interventions: Drug: ASC-J9
- 0.1% ASC-J9 cream (Experimental)
  Interventions: Drug: ASC-J9

INTERVENTIONS:
Drug: ASC-J9 — Cream for twice daily topical application to the face

SUMMARY:
To evaluate the safety and efficacy of topical 0.1% and 0.025% ASC-J9 creams applied twice daily for facial acne compared to vehicle control.

DETAILED DESCRIPTION:
Approximately 180 patients at least 12 years of age with facial acne will be randomized to twice daily topical treatment with 0.1% or 0.025% ASC-J9 cream or vehicle control for 12 weeks. Patients will return to the clinic at Weeks 2, 4, 8 and 12 and again 4 weeks after the last dose of study drug for evaluation of acne status and safety parameters.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 12 years of age at the time of enrollment
* Facial acne, with:

  1. 20-60 inflammatory facial lesions (papules/pustules/nodules/cysts);
  2. 20-100 noninflammatory facial lesions (open and closed comedones);
  3. No more than 2 nodules/cysts on the face (defined as an inflammatory lesion greater than or equal to 5 mm in diameter);
  4. Investigator's Global Assessment (IGA) acne score of 3 or 4.

Key Exclusion Criteria:

* Females who are pregnant or breast-feeding
* Skin diseases other than acne vulgaris
* Use of other topical or systemic treatments for acne
* Other significant medical conditions or clinically significant abnormal laboratory test results.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Dosik, MD, Principal Investigator — TKL Research; Chieh-Chen Huang, MD, Principal Investigator — Shih Kong Wu Ho-Su Memorial Hospital; Chih-Hsun Yang, MD, Principal Investigator — Chang Gung Memorial Hospital; Ting-Jui Chen, MD, Principal Investigator — Wan Fang Hospital; Wei-Ming Wang, MD PhD, Principal Investigator — Tri-Service General Hospital; Kuo-Hsien Wang, MD, Principal Investigator — Taipei Medical University Hospital; Ji-Chen Ho, MD, Principal Investigator — Chang Gung Memorial Hospital Kaohsiung Branch
Locations (7):
- TKL Research, Inc, Paramus, New Jersey, United States
- Taiwan (6):
  - Chang Gung Memorial Hospital, NiaoSong District, Kaohsiung City
  - Shih Kong Wu Ho-Su Memorial Hospital, Taipei City, Taipei
  - Tri-Service General Hospital, Taipei City, Taipei
  - Taipei Medical University Hospital, Taipei City, Taipei
  - Wan Fang Hospital, Taipei, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Gueishan Township, Taoyuan County

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Control Cream | 0.025% ASC-J9 Cream | 0.1% ASC-J9 Cream
Started | 58 | 60 | 63
Completed | 51 | 57 | 60
Not Completed | 7 | 3 | 3
Not completed — Lack of Efficacy | 4 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Subject wanted alternate treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Control Cream | 0.025% ASC-J9 Cream | 0.1% ASC-J9 Cream | Total
Number analyzed (Participants) | 58 | 60 | 63 | 181
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.1 (5.7) | 20.7 (4.8) | 22.0 (6.3) | 21.3 (5.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 18 | 22 | 58
  Between 18 and 65 years | 40 | 42 | 41 | 123
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 32 | 86
  Male | 27 | 37 | 31 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 44 | 48 | 49 | 141
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4
  White | 14 | 10 | 11 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 56 | 58 | 62 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 15 | 42
  Taiwan | 44 | 47 | 48 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Inflammatory Acne Lesion Counts
Description: Percent change from Baseline
Time Frame: 12 weeks
Population: All randomized patients
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Groups:
- Vehicle Control Cream: Vehicle control cream for twice daily topical application to the face
Arm/Group | Vehicle Control Cream | 0.025% ASC-J9 Cream | 0.1% ASC-J9 Cream
Number analyzed (Participants) | 58 | 60 | 63
Percentage change from baseline | -28.6 (52.2) | -44.3 (31.7) | -44.4 (34.6)
Statistical Analysis 1: Comparison: Vehicle Control Cream vs 0.025% ASC-J9 Cream vs 0.1% ASC-J9 Cream; Test type: Superiority or Other; p = 0.1919, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) row mean score statistics, adjusting for investigational site

2. Secondary Outcome: Success on Investigator Global Assessment (IGA) at Week 12
Description: Overall acne rated as clear, almost clear, mild, moderate, severe, very severe.
  Success = Week 12 rating of clear or almost clear and at least a 2-grade improvement from baseline
Time Frame: 12 weeks
Population: All randomized subjects
Measure: Number; unit: Percentage of subjects
Arm/Group | Vehicle Control Cream | 0.025% ASC-J9 Cream | 0.1% ASC-J9 Cream
Number analyzed (Participants) | 58 | 60 | 63
Percentage of subjects | 6.9 | 21.7 | 17.5
Statistical Analysis 1: Comparison: Vehicle Control Cream vs 0.025% ASC-J9 Cream vs 0.1% ASC-J9 Cream; Test type: Superiority or Other; p = 0.0610, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent Change in Noninflammatory Acne Lesion Counts
Description: Percent change from Baseline
Time Frame: 12 weeks
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Vehicle Control Cream | 0.025% ASC-J9 Cream | 0.1% ASC-J9 Cream
Number analyzed (Participants) | 58 | 60 | 63
Percentage change from baseline | -18.5 (49.7) | -35.5 (39.7) | -36.3 (38.6)
Statistical Analysis 1: Comparison: Vehicle Control Cream vs 0.025% ASC-J9 Cream vs 0.1% ASC-J9 Cream; Test type: Superiority or Other; p = 0.0857, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: During 12-week dosing period and for 4 weeks after the last dose.
Arm/Group | Vehicle Control Cream | 0.025% ASC-J9 Cream | 0.1% ASC-J9 Cream
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 0/58 | 0/60 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No